CLINICAL TRIAL: NCT05514509
Title: A Phase 4, Randomized, Open-label, Three-arm Study to Evaluate Implementation Strategies for the Delivery of CAB for HIV Pre-exposure Prophylaxis (PrEP) Across Clinical Settings for Adult (≥18 Years) Black cis-and Transgender Women Without HIV Infection Living in the United States Ending the Epidemic (EHE) Territories
Brief Title: A Study Evaluating Implementation Strategies for the Delivery of APRETUDE for Black cis-and Transgender Women in United States EHE Territories
Acronym: EBONI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 217711
Expanded Access: NCT03462810 (Available)
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: HIV Infections
Keywords: Cabotegravir; Long acting injectables; Implementation science; HIV; PrEP; HIV Disparities; Ending the Epidemic; Engaging Black Women on APRETUDE by Optimizing Novel Implementation Strategies (EBONI)
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Standard Implementation (SI) (Active Comparator): PSPs will receive APRETUDE injection and could receive optional Cabotegravir tablets as oral lead in (OLI). The SI arm receives the standard toolkits that are anticipated to be available for APRETUDE that includes information resource for PSPs and SSPs.
  Interventions: Drug: APRETUDE; Drug: Cabotegravir tablet
- Enhanced Implementation (EI) (Experimental): PSPs will receive APRETUDE injection and could receive optional Cabotegravir tablets as OLI. The EI arm will receive all components of SI arm and additional provider-focused implementation strategies. Provider-focused strategies will include a patient-provider communication tool, Provider Education, and enhanced tool kit materials.
  Interventions: Drug: APRETUDE; Drug: Cabotegravir tablet
- Enhanced Collaborative Implementation (ECI) (Experimental): PSPs will receive APRETUDE injection and could receive optional Cabotegravir tablets as OLI. The ECI arm will involve implementation strategies to support patient activation and provider awareness. Clinics randomized to ECI will receive all components of SI and additional implementation strategies to support patient activation and ensure provider awareness. ECI strategies will include a patient information and product resources and peer support.
  Interventions: Drug: APRETUDE; Drug: Cabotegravir tablet

INTERVENTIONS:
Drug: APRETUDE — Available as intramuscular injection.
Drug: Cabotegravir tablet — Available as marketed orally administered tablets.

SUMMARY:
The purpose of the study is to evaluate the appropriateness, adoption, feasibility, fidelity, and acceptability of implementation strategies and Cabotegravir (CAB) pre-exposure prophylaxis (PrEP). The study objectives are also to identify barriers and facilitators to implementation. The first of two participant types in the study are the Patient Study Participants (PSPs) will refer to individuals who are enrolled in the study and who will receive commercially available CAB PrEP via prescription from the PrEP provider. The second are Staff Study Participants (SSPs) who are site staff involved in the administrative and clinical aspects of offering and administering PrEP to PSPs at the clinical site.

ELIGIBILITY:
Inclusion criteria:

* Participant must be ≥18 years of age, at the time of signing the informed consent.
* HIV negative at screening. Type of HIV-1 test is per standard of care.
* No prior history of receiving oral CAB or CAB LA injections.
* PrEP provider deems CAB PrEP use to be appropriate per the applicable CAB PrEP prescribing information prior to enrollment in the study.
* Female at birth or self-identified Transgender Female.
* Self-identified as African American/Black
* Capable of giving signed informed consent

Exclusion criteria:

* HIV indeterminate or positive test result during screening.
* A participant of concurrent interventional clinical or implementation science study at any time during the study.
* Cis-gender or Transgender male

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female at birth or self-identified Transgender Female
Enrollment: 370 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2025-09-02 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Mean Intervention Appropriateness Measure (IAM) Score in SSPs | Up to Month 13
  The responses for appropriateness will be measured on a Likert scale ranging from 0 to 5 with higher values representing better outcomes.

SECONDARY OUTCOMES:
Mean IAM Score in SSPs at Month 1, 4, 5, 12 and 13 | Month 1, 4, 5, 12 and 13
  The responses for appropriateness will be measured on a Likert scale ranging from 0 to 5 with higher values representing better outcomes. Data will be collected at Month 1, 4, and 12 for participants who start with injections and at Month 1, 5, 13 for participants who start with the oral lead in.
Change from Baseline in Mean IAM Score in SSPs at Month 4, 5, 12 and 13 | Baseline (Month 1) and Month 4, 5, 12 and 13
  The responses for appropriateness will be measured on a Likert scale ranging from 0 to 5 with higher values representing better outcomes. Data will be collected at Month 1, 4, and 12 for participants who start with injections and at Month 1, 5, 13 for participants who start with the oral lead in.
Appropriateness of APRETUDE Assessed by SSP Questionnaire responses at Month 1, 4, 5, 12 and 13 | Month 1, 4, 5, 12 and 13
  Data will be collected at Month 1, 4, and 12 for participants who start with injections and at Month 1, 5, 13 for participants who start with the oral lead in.
Appropriateness of APRETUDE Assessed by Semi-structured interview (SSI) at Month 4, 5, 12 and 13 | Month 1, 4, 5, 12 and 13
  Appropriateness of APRETUDE will be measured from themes emerging from Proctor and Consolidated Framework for Implementation Research (CFIR) guided semi-structured qualitative interview. Data will be collected at Month 1, 4, and 12 for participants who start with injections and at Month 1, 5, 13 for participants who start with the oral lead in.
Appropriateness of APRETUDE Assessed by Semi-structured interview (SSI) at Month 4, 5, 12 and 13 | Month 4, 5 12 and 13
  Appropriateness of APRETUDE will be measured from themes emerging from Proctor and CFIR framework guided semi-structured qualitative interview. Data will be collected at Month 4, and 12 for participants who start with injections and at Month 5, 13 for participants who start with the oral lead in.
Mean IAM Score in PSPs at Month 1, 4, 5, 12 and 13 | Month 1, 4, 5, 12 and 13
  The responses for appropriateness will be measured on a Likert scale ranging from 0 to 5 with higher values representing better outcomes. Data will be collected at Month 1, 4, and 12 for participants who start with injections and at Month 1, 5, 13 for participants who start with the oral lead in.
Change from Baseline in Mean IAM Score in PSPs at Month 4, 5, 12 and 13 | Baseline (Month 1) and Month 4, 5, 12 and 13
  The responses for appropriateness will be measured on a Likert scale ranging from 0 to 5 with higher values representing better outcomes. Data will be collected at Month 1, 4, and 12 for participants who start with injections and at Month 1, 5, 13 for participants who start with the oral lead in.
Perception of Appropriateness of APRETUDE Assessed by PSP Questionnaire responses at Month 1, 4, 5, 12 and 13 | Month 1, 4, 5, 12 and 13
  Data will be collected at Month 1, 4, and 12 for participants who start with injections and at Month 1, 5, 13 for participants who start with the oral lead in.
Perception of Appropriateness of APRETUDE Assessed by SSI in PSPs at Month 4, 5, 12 and 13 | Month 4, 5, 12 and 13
  Perception of Appropriateness of APRETUDE will be measured from themes emerging from Proctor and CFIR framework guided semi-structured qualitative interview. Data will be collected at Month 4, and 12 for participants who start with injections and at Month 5, 13 for participants who start with the oral lead in.
Number of cis-and trans Black women who Complete a Sexual Health Assessment through Month 13 in ECI Arm based on site-level PrEP Information Questionnaire | Up to Month 13
Number of PSPs who Complete a Sexual Health Assessment through Month 13 in ECI Arm based on Site-level PrEP Information Questionnaire | Up to Month 13
Number of cis-and trans Black Women who Initiate APRETUDE through Month 13 by Study Arm Based on Site level PrEP Information Questionnaire | Up to Month 13
Number of cis-and trans Black Women who Initiate APRETUDE through Month 13 by Clinic Characteristics Based on Site level PrEP Information Questionnaire | Up to Month 13
Proportion of cis-and trans Black Women who Initiate APRETUDE through Month 13 by Study Arm Based on Site level PrEP Information Questionnaire | Up to Month 13
Proportion of cis-and trans Black Women who Initiate APRETUDE through Month 13 by Clinic Characteristics Based on Site level PrEP Information Questionnaire | Up to Month 13
Number of cis-and trans Black Women who Continue APRETUDE beyond a First Dose through Month 13 by study arm based on Site-level PrEP Information Questionnaire | Up to Month 13
Number of cis-and trans Black Women who Continue APRETUDE beyond a First Dose through Month 13 by Clinic Characteristics based on Site-level PrEP Information Questionnaire | Up to Month 13
Mean Feasibility of Intervention Measure (FIM) score in SSPs for Implementation Strategies | Month 1 and 4, 5, 12 and 13
  The responses for feasibility will be measured on a 5-point Likert scale ranging from 0 to 5 with higher values representing better outcomes. Data will be collected at Month 1, 4, and 12 for participants who start with injections and at Month 1, 5, 13 for participants who start with the oral lead in.
Change from Baseline in FIM Score in SSPs for Implementation Strategies | Baseline (Month 1) and Month 4, 5, 12 and 13
  The responses for feasibility will be measured on a 5-point Likert scale ranging from 0 to 5 with higher values representing better outcomes. Data will be collected at Month 1, 4, and 12 for participants who start with injections and at Month 1, 5, 13 for participants who start with the oral lead in.
Feasibility of Strategy Assessed by SSPs Questionnaire responses at Month 1, 4, 5, 12 and 13 | Month 1, 4, 5, 12 and 13
  Data will be collected at Month 1, 4, and 12 for participants who start with injections and at Month 1, 5, 13 for participants who start with the oral lead in.
Feasibility and Utility of Strategy Assessed in SSPs by SSI at Month 4, 5, 12 and 13 | Month 4, 5, 12 and 13
  Perception of Appropriateness of APRETUDE will be measured from themes emerging from Proctor and CFIR framework guided semi-structured qualitative interview. Data will be collected at Month 4, and 12 for participants who start with injections and at Month 5, 13 for participants who start with the oral lead in.
Proportion of SSPs that Respond in Agreement on Relevant Items on the Implementation science questionnaire (ISQ) that each implementation tool and strategy is fit for use through Month 13 Based on Study Arm | Up to Month 13
  ISQ measures a range, including acceptability, feasibility, and utility.
Proportion of SSPs that Respond in Agreement on Relevant Items on the ISQ that each implementation tool and strategy is fit for use through Month 13 Based on Clinic Characteristics | Up to Month 13
  ISQ measures a range, including acceptability, feasibility, and utility.
Proportion of SSPs that Respond in Agreement on Relevant Items on the ISQ that each implementation tool and strategy is fit for use through Month 13 Based on Patient Subgroups | Up to Month 13
  ISQ measures a range, including acceptability, feasibility, and utility.
Proportion of PSPs that Respond in Agreement on Relevant Items on the Implementation science questionnaire (ISQ) that each implementation tool and strategy is fit for use through Month 13 Based on Study Arm | Up to Month 13
  ISQ measures a range, including acceptability, feasibility, and utility.
Proportion of PSPs that Respond in Agreement on Relevant Items on the ISQ that each implementation tool and strategy is fit for use through Month 13 Based on Clinic Characteristics | Up to Month 13
  ISQ measures a range, including acceptability, feasibility, and utility.
Proportion of PSPs that Respond in Agreement on Relevant Items on the ISQ that each implementation tool and strategy is fit for use through Month 13 Based on Patient Subgroups | Up to Month 13
  ISQ measures a range, including acceptability, feasibility, and utility.
Perceptions of Utility of Implementation tools and strategies Assessed by SSIs in PSPs through Month 13 based on Patient Subgroups | Up to Month 13
  Perceptions of Utility of Implementation tools and strategies will be measured from themes emerging from Proctor and CFIR framework guided semi-structured qualitative interview.
Proportion of Injections Occurring Within Target Window from Target Date (+-7 days of target date) | Up to Month 13
Perception of Barriers and Facilitators to Fidelity to Injections Window Assessed by SSIs in PSPs | Month 1, 12 and 13
  Perception of Barriers and Facilitators to Fidelity to Injections Window will be measured from themes emerging from Proctor and CFIR framework guided semi-structured qualitative interview. Data will be collected at Month 1 and 12 for participants who start with injections and at Month 1 and 13 who start with oral lead in.
Perception of Barriers and Facilitators to Fidelity to Injections Window Assessed by Surveys in PSPs | Month 1, 4, 5, 12 and 13
  Data will be collected at Month 1, 4, and 12 for participants who start with injections and at Month 1, 5, 13 for participants who start with the oral lead in.
Perception of Barriers and Facilitators to Fidelity to Injections Window Assessed by Implementation Monitoring Calls (IMC) in SSPs | Month 4, 5, 12 and 13
  Data will be collected at Month 4, and 12 for participants who start with injections and at Month 5 and 13 for participants who start with the oral lead in.
Proportion of PSPs completing target number of injections | Up to Month 13
Barriers, Facilitators, Concerns and Perception to Implementation in SSPs and PSPs Assessed by Questionnaire responses | Month 1, 4, 5, 12 and 13
  Data will be collected at Month 1, 4, and 12 for participants who start with injections and at Month 1, 5, 13 for participants who start with the oral lead in.
Perception to Facilitators and Barriers to Implementation in SSPs Assessed by SSI | Month 4, 5, 12 and 13
  Perception to Facilitators and Barriers to Implementation will be measured from themes emerging from Proctor and CFIR framework guided semi-structured qualitative interview. Data will be collected at Month 4, and 12 for participants who start with injections and at Month 5 and 13 for participants who start with the oral lead in.
Perception to Facilitators and Barriers to Implementation in SSPs Assessed by IMC | Month 4, 5, 12 and 13
  Data will be collected at Month 4, and 12 for participants who start with injections and at Month 5 and 13 for participants who start with the oral lead in.
Perception to Facilitators and Barriers to Implementation in PSPs Assessed by SSI | Month 1, 12 and 13
  Perception to Facilitators and Barriers to Implementation will be measured from themes emerging from Proctor and CFIR framework guided semi-structured qualitative interview. Data will be collected at Month 1 and 12 for participants who start with injections and at Month 1 and 13 for participants who start with the oral lead in.
Acceptability of Intervention Measure (AIM) Score for APRETUDE in SSPs and PSPs | Month 1, 4, 5, 12 and 13
  The responses for acceptability will be measured on a Likert scale ranging from 0 to 5 with higher values representing better outcomes. Data will be collected at Month 1, 4, and 12 for participants who start with injections and at Month 1, 5, 13 for participants who start with the oral lead in.
FIM Score for APRETUDE in SSPs and PSPs | Month 1, 4, 5, 12 and 13
  The responses for feasibility will be measured on a Likert scale ranging from 0 to 5 with higher values representing better outcomes. Data will be collected at Month 1, 4, and 12 for participants who start with injections and at Month 1, 5, 13 for participants who start with the oral lead in.
Feasibility and Acceptability of APRETUDE in SSPs and PSPs Assessed by Questionnaire Responses | Month 1, 4, 5, 12 and 13
  Data will be collected at Month 1, 4, and 12 for participants who start with injections and at Month 1, 5, 13 for participants who start with the oral lead in.
Feasibility and Acceptability of APRETUDE in SSPs Assessed by SSIs | Month 4, 12 and 13
  Feasibility and Acceptability of APRETUDE will be measured from themes emerging from Proctor and CFIR framework guided semi-structured qualitative interview. Data will be collected at Month 4, and 12 for participants who start with injections and at Month 13 for participants who start with the oral lead in.
Feasibility and Acceptability of APRETUDE in PSPs Assessed by SSIs | Month 1, 12 and 13
  Feasibility and Acceptability of APRETUDE will be measured from themes emerging from Proctor and CFIR framework guided semi-structured qualitative interview. Data will be collected at Month 1 and 12 for participants who start with injections and at Month 1 and 13 for participants who start with the oral lead in.
Proportion of PSPs that have one Oral lead-in before CAB Injection | Up to Month 13
Perception on Reason for Decision to Use Oral lead-in in SSPs Assessed by SSI | Month 1, 4, 5, 12 and 13
  Perception on Reason for Decision to Use Oral lead-in will be measured from themes emerging from Proctor and CFIR framework guided semi-structured qualitative interview. Data will be collected at Month 1, 4, and 12 for participants who start with injections and at Month 1, 5, 13 for participants who start with the oral lead in.
Perception on Reason for Decision to Use Oral lead-in SSPs Assessed by Survey responses | Month 1, 4, 5, 12 and 13
  Data will be collected at Month 1, 4, and 12 for participants who start with injections and at Month 1, 5, 13 for participants who start with the oral lead in.
Perception on Reason for Decision to Use Oral lead-in PSPs Assessed by SSIs | Month 1
  Perception on Reason for Decision to Use Oral lead-in will be measured from themes emerging from Proctor and CFIR framework guided semi-structured qualitative interview.
Perception on Reason for Decision to Use Oral lead-in PSPs Assessed by Survey Responses | Month 1
Proportion of PSPs that Complete a Sexual Health Assessment and Start or Switch from Oral PrEP to APRETUDE | Up to Month 13
Reasons for Choosing or Switching from Oral PrEP to APRETUDE in PSPs Assessed by SSIs | Up to Month 13
  Reasons for Choosing or Switching from Oral PrEP to APRETUDE will be measured from themes emerging from Proctor and CFIR framework guided semi-structured qualitative interview.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (16):
- United States (16):
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Bridgeport, Kansas
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

REFERENCES:
- [Derived] Nelson KL, Evans Cooper T, Lawson Y, Baker D, Mocherla S, Dieterich M, Hodge T, Dyson A, Sutherland-Philips D, Swygard H, Petty L, Jeffery P, Sutton K, Bonner CP, Andrews SM, Chang S, Budnik P, Smith K, de Ruiter A, Czarnogorski M, Pilgrim N. Strategies for implementing long-acting cabotegravir for PrEP in US clinics serving Black women: interim healthcare provider findings from the EBONI study. J Int AIDS Soc. 2025 Jul;28 Suppl 2(Suppl 2):e26497. doi: 10.1002/jia2.26497. PMID 40600480